CLINICAL TRIAL: NCT01132794
Title: A Study to Assess the Analgesia and Sedation Using Intranasal Dexmedetomidine in Third Molar Surgery Under Local Anaesthesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Other Study IDs: 200707176037
Record Dates: First submitted 2010-05-24; First posted 2010-05-28 (Estimated); Last update posted 2010-06-16 (Estimated); Status verified 2010-05

CONDITIONS: Pain; Sedation
Keywords: Pain relief and sedation condition
MeSH Terms: conditions — Pain

ARMS (2):
- Placebo (Placebo Comparator): Intranasal nasal saline
  Interventions: Drug: Placebo
- Dexmedetomidine (Active Comparator): Intranasal dexmedetomidine
  Interventions: Drug: Intranasal dexmedetomidine

INTERVENTIONS:
Drug: Intranasal dexmedetomidine — 1mcg per kg dexmedetomidine given intranasally 45 minutes before operation
  Arms: Dexmedetomidine
Drug: Placebo — Intranasal nasal saline
  Arms: Placebo

SUMMARY:
Dental procedures such as wisdom tooth removal evoke very high levels of patients' anxiety and it is, therefore, common practice to provide concomitant pharmacologic sedation.

Sedative agents can be administered by the oral, rectal, intra muscular and intravenous routes. The oldest, safest and most convenient route at present is the oral route. However, as Uygur-Bayramicli et al. mentioned that administering the drugs orally can result in problems like delayed effect. Intranasal administration is a straightforward procedure. It is simple and relatively painless. Although it may be objectionable, less patient cooperation is required than with oral administration, especially in which the child must swallow the medication.

Many studies on dental sedation have been carried out by anesthesiologists but there is no ideal drug that can offer effects of both sedation and analgesia. Some drugs offer only one effect and others are not safe enough for clinical use. Midazolam, a benzodiazepine drug, is the traditional choice for sedation, but it has properties such as relatively slow onset and no analgesia. Propofol is an alkylphenol sedative and hypnotic agent with a rapid onset and offset. It has been used in patient controlled sedation before. But it has no analgesic properties. It can provide some antegrade amnesia, but it is not as reliable an amnestic as the benzodiazepine drugs. Because of these characteristics, propofol often is supplemented with narcotics and benzodiazepines. Although not irritant, it can cause pain during intravenous infusion.

A new drug, an alpha agonist with its relatively high ratio of α2/α1-activity (1620:1 as compared with 220:1 for clonidine) of theα2 receptor is dexmedetomidine. This property may lead to more potent effects of both sedation and analgesia without unwanted cardiovascular effects fromα1 receptor activation. Most of the data evaluating the use of dexmedetomidine in the intensive care unit (ICU) were obtained in the immediate postoperative period, mainly in patients who underwent open-heart surgery. Currently, clinicians are awaiting studies in broader patient populations. In the studies that have been completed to date, sedation has been attained easily with maintenance of respiratory function. Patients are readily arousable. There is a minimal increase in blood pressure initially, followed by a slight decrease in blood pressure. Lower dose ranges, avoidance of rapid bolus injection, and a slow rate of administration tend to decrease these circulatory side effects. So many clinical studies have shown that it can be well and safely used intravenously, intramuscularly and transdermally. Although not an officially technique, there are also reports of intranasal administration resulting in fairly predictable onset in both adults and children.

The investigators propose that intranasal can help to improve postoperative pain relief with better sedation.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) 1 or 2
* Age >18 and less than 40 years
* Unilateral wisdom tooth removal
* Written informed consent

Exclusion Criteria:

* Allergy to dexmedetomidine and propofol
* Patient refusal
* Mentally unfit
* Impaired renal or hepatic function
* Pregnant
* Exposure to study drug within the past 3 months.
* Use ofα2 agonists currently
* Patients with cardiac disease
* Abnormal electrocardiogram
* Inability to complete psychomotor test
* Addictive in illicit drugs or alcohol

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult

PRIMARY OUTCOMES:
Pain scores after operation

SECONDARY OUTCOMES:
Sedation satisfaction

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, The University of Hong Kong, Hong Kong, Hong Kong